CLINICAL TRIAL: NCT06411288
Title: A Phase 3 Randomized, Double-Blind, Placebo-Controlled, Global Study to Evaluate the Efficacy and Safety of Intravenous AOC 1001 for the Treatment of Myotonic Dystrophy Type 1
Brief Title: Global Study of Del-desiran for the Treatment of DM1
Acronym: HARBOR
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Avidity Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AOC 1001-CS3
Record Dates: First submitted 2024-05-08; First posted 2024-05-13 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: DM1; Myotonic Dystrophy; Myotonic Dystrophy 1; Myotonia; Myotonic Dystrophy Type 1 (DM1); Dystrophy Myotonic; Myotonic Disorders; Steinert Disease; Steinert; Myotonic Muscular Dystrophy
Keywords: DM1; Myotonic Dystrophy; Myotonic Dystrophy 1; Myotonia; Myotonic Dystrophy Type 1 (DM1); Dystrophy Myotonic; Myotonic Disorders; Steinert Disease; Steinert; Myotonic Muscular Dystrophy; HARBOR; Avidity Biosciences; Avidity; AOC 1001; Del-desiran; Delpacibart etedesiran
MeSH Terms: conditions — Myotonic Dystrophy; Myotonia; Myotonic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Del-desiran (Experimental): Del-desiran (AOC 1001) will be administered seven times
  Interventions: Drug: AOC 1001 (del-desiran)
- Placebo (Placebo Comparator): Saline will be administered seven times
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AOC 1001 (del-desiran) — Del-desiran will be administered by intravenous (IV) infusion.
  Arms: Del-desiran
Drug: Placebo — Placebo will be administered by intravenous (IV) infusion.
  Arms: Placebo

SUMMARY:
A Phase 3 Randomized, Double-Blind, Placebo-Controlled, Global Study to Evaluate the Efficacy and Safety of Intravenous Delpacibart Etedesiran (abbreviated del-desiran, formerly AOC 1001) for the Treatment of Myotonic Dystrophy Type 1

DETAILED DESCRIPTION:
The study consists of a Screening Period of up to 6 weeks and 54-week Treatment Period. The anticipated duration is approximately 60 weeks.

Participants will be randomized to receive an intravenous infusion of either del-desiran or placebo at the clinical study site every 8 weeks for a total of 7 doses. The final dose will occur at Week 48, followed by a final assessment at Week 54.

After completion of Week 54 assessments, eligible participants will have the option to enroll into an open label extension (OLE) study, pending regulatory approval.

An Independent Data Monitoring Committee (IDMC) comprised of members independent and external to the Sponsor will review safety, tolerability, and efficacy (as needed) data of this study at regular intervals.

ELIGIBILITY:
Key Inclusion Criteria:

* Clinical and genetic diagnosis (CTG repeat ≥ 100) of DM1
* Ability to walk independently (orthoses and ankle braces allowed) for at least 10 meters at screening

Key Exclusion Criteria:

* Breastfeeding, pregnancy, or intent to become pregnant during the study
* Unwilling or unable to comply with contraceptive requirements
* Abnormal lab values, conditions or diseases that would make the participant unsuitable for the study
* Diabetes that is not adequately controlled
* History of decompensated heart failure within 3 months of screening. Participants with preexisting pacemaker/ICD are not excluded.
* Body Mass Index > 35 kg/m2 at Screening
* Recently treated with an investigational drug or biological agent
* Treatment with anti-myotonic medication within 5 half-lives or 14 days of baseline, whichever is longer, prior to baseline.

Note: Additional protocol defined Inclusion and Exclusion criteria apply

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Hand function | Through Week 54
  video Hand Opening Time (vHOT)

SECONDARY OUTCOMES:
Hand grip strength | Through Week 54
  by dynamometer
Quantitative Muscle Testing composite score | Through Week 54
  by dynamometer
Myotonic Dystrophy Type 1 activity and participation scale c | Through Week 54
10-Meter Walk/Run Test | Through Week 54
  Time (in seconds) to walk or run 10 meters

CONTACTS AND LOCATIONS:
Locations (34):
- United States (18):
  - Stanford University, Stanford, California
  - University of Colorado, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - University Research Center of South Florida, Tampa, Florida
  - Indiana University (IU), Indianapolis, Indiana
  - Kansas University Medical Center, Kansas City, Kansas
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - University of Rochester Medical Center, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest, Winston-Salem, North Carolina
  - University of Cincinnati Gardner Neuroscience Institute, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Houston Methodist Neurological Institute, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington, Seattle, Washington
- Canada (2):
  - The Ottawa Hospital, Ottawa, Ontario
  - Montreal Neurological Institute, Montreal, Quebec
- Denmark (2):
  - Aarhus University Hospital, Aarhus N
  - Rigshospitalet, Copenhagen
- AP-HP Hopital Pitie-Salpetriere, Paris, France
- Klinikum der Ludwig-Maximilians-Universitaet Muenchen, Munich, Germany
- Fondazione Serena Onlus - Centro Clinico NeMO Milano, Milan, Italy
- Japan (4):
  - Aomori Hospital, Aomori, Aomori
  - National Hospital Organization Osaka Toneyama Medical Center, Osaka
  - Osaka University Hospital, Osaka
  - National Center of Neurology and Psychiatry, Tokyo
- Netherlands (2):
  - Maastricht University Medical Center, Maastricht
  - Stichting Radboud Universitair Medisch Centrum, Nijmegen
- Hospital Universitario Donostia, Donostia / San Sebastian, Spain
- United Kingdom (2):
  - University College London Hospital, London
  - St. Georges University Hospitals NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Undecided